CLINICAL TRIAL: NCT05610943
Title: Comparison of The Postoperative Analgesic Effectiveness of Ultrasound-Guided Quadratus Lumborum Block and Ilioinguinal Iliohypogastric Nerve Block in Pediatric Inguinal Hernia Operation, Prospective Randomized Controlled Study
Brief Title: Comparison of The Quadratus Lumborum Block and Ilioinguinal Iliohypogastric Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Altınay, principal investigator, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2977
Record Dates: First submitted 2022-10-28; First posted 2022-11-09 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Post Operative Pain; Inguinal Hernia; Quadratus Lumborum Nerve Block
Keywords: quadratus lumborum nerve block; postoperative pain; inguinal herniae; ilio-inguinal iliohypogastric nerve block
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- quadratus lumborum nerve block (Active Comparator): In Group Q; The patient was placed in the lateral position with the side to be blocked on top. After providing skin antisepsis with 5% povidone iodine, sterile dressing was applied. After the USG probe was covered with a sterile sheath, it was placed transversely between the iliac crest and the costa edge. After imaging the external-internal oblique and transversus abdominis muscles, the probe was advanced posteriorly. Quadratus lumborum, Psoas Major and Erector Spina muscles were visualized. The needle was advanced towards the middle thoracolumbar fascia between the Quadratus lumborum muscle and the Erector Spina muscle with the in-plane technique, and the location was confirmed by injecting 1 ml of 0.9 saline. 0.25% Bupivacaine was injected at a dose of 0.5 mL/kg after negative aspiration.
  Interventions: Procedure: ultrasound-guided quadratus lumborum nerve block
- Ilioinguinal Iliohypogastric Nerve Block (Active Comparator): In Group I; The patient was placed in the supine position. After providing skin antisepsis with 5% povidone iodine, sterile dressing was applied. After the USG probe was covered with a sterile sheath, it was placed on the anterior abdominal wall parallel to the imaginary line between the umbilicus and the anterior superior iliac wing. After imaging the external-internal oblique and transversus abdominis muscles, the ilioinguinal-iliohypogastric nerve was visualized as two small hypoechoic areas between the internal oblique muscle and the transversus abdominis muscle. The location was confirmed by injecting 1 ml of 0.9 saline by advancing the needle with the in-plane technique close to the nerve structures. 0.25% Bupivacaine was injected at a dose of 0.5 mL/kg after negative aspiration.
  Interventions: Procedure: ultrasound-guided Ilioinguinal Iliohypogastric Nerve Block

INTERVENTIONS:
Procedure: ultrasound-guided quadratus lumborum nerve block — The patient was placed in the lateral position with the side to be blocked on top. After providing skin antisepsis with 5% povidone iodine, sterile dressing was applied. After the USG probe was covered with a sterile sheath, it was placed transversely between the iliac crest and the costa edge. After imaging the external-internal oblique and transversus abdominis muscles, the probe was advanced posteriorly. Quadratus lumborum, Psoas Major and Erector Spina muscles were visualized. The needle was advanced towards the middle thoracolumbar fascia between the Quadratus lumborum muscle and the Erector Spina muscle with the in-plane technique, and the location was confirmed by injecting 1 ml of 0.9 saline. 0.25% Bupivacaine was injected at a dose of 0.5 mL/kg after negative aspiration.
  Arms: quadratus lumborum nerve block
Procedure: ultrasound-guided Ilioinguinal Iliohypogastric Nerve Block — The patient was placed in the supine position. After providing skin antisepsis with 5% povidone iodine, sterile dressing was applied. After the USG probe was covered with a sterile sheath, it was placed on the anterior abdominal wall parallel to the imaginary line between the umbilicus and the anterior superior iliac wing. After imaging the external-internal oblique and transversus abdominis muscles, the ilioinguinal-iliohypogastric nerve was visualized as two small hypoechoic areas between the internal oblique muscle and the transversus abdominis muscle. The location was confirmed by injecting 1 ml of 0.9 saline by advancing the needle with the in-plane technique close to the nerve structures. 0.25% Bupivacaine was injected at a dose of 0.5 mL/kg after negative aspiration.
  Arms: Ilioinguinal Iliohypogastric Nerve Block

SUMMARY:
Perioperative and postoperative pain control in pediatric patients is a frequently neglected issue. Regional anesthesia applications reduce adverse drug events by minimizing opioid consumption and provide effective and safe analgesia. In recent years, quadratus lumborum block has emerged as an alternative regional anesthesia technique and it has been shown to provide analgesia as effectively as caudal block in children, and in a limited number of studies it has been said that it is more effective than transversus abdominis plane block. There are few studies in the literature comparing ilioinguinal iliohypogastic nerve block and quadratus lumborum block in children.

DETAILED DESCRIPTION:
Perioperative and postoperative pain control in pediatric patients is a frequently neglected issue. Providing effective perioperative analgesia reduces surgical stress, making the postoperative period more comfortable both physiologically and psychologically, effective postoperative pain control reduces the length of stay in the hospital, and also contributes to the long-term positive personality development of children.

Physiological, pharmacokinetic and pharmacodynamic differences in children delay the metabolism and excretion of systemic analgesics, resulting in a prolonged effect and an increased risk of apnea. Regional anesthesia applications reduce adverse drug events by minimizing opioid consumption and provide effective and safe analgesia.

Caudal block, which is a common regional anesthesia practice in inguinal hernia surgery in children, has disadvantages such as motor block and urinary retention. With the introduction of ultrasonography, peripheral block techniques such as transversus abdominis plane block and ilioinguinal iliohypogastric nerve block have been shown to provide effective and safe analgesia and have replaced central blocks. In recent years, quadratus lumborum block has emerged as an alternative regional anesthesia technique and it has been shown to provide analgesia as effectively as caudal block in children, and in a limited number of studies it has been said that it is more effective than transversus abdominis plane block. There are few studies in the literature comparing ilioinguinal iliohypogastric nerve block and quadratus lumborum block in children.

The purpose of the study to compare the postoperative analgesic effectiveness of quadratus lumborum block and ilioinguinal iliohypogastric block in pediatric patients who underwent unilateral inguinal hernia operation.

ELIGIBILITY:
Inclusion Criteria:

* who were scheduled for unilateral inguinal hernia operation
* with American Society of Anesthesiologists (ASA) physical score I-II
* aged 2-7 years

Exclusion Criteria:

* Patients with coagulopathy
* skin infection at the block application site
* bupivacaine allergy
* neuropsychiatric disease

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
FLACC score | 24 hours
  Face, Legs, Activity, Cry, Consolability (FLACC) Behavioral Pain Scale. FLACC is a behavioral pain assessment scale used for nonverbal or preverbal patients who are unable to self-report their level of pain. Pain is assessed through observation of 5 categories including face, legs, activity, cry, and consolability. The increase in the pain felt by the patient also increases the flacc score. Each category is scored on the 0-2 scale which results in a total score of 0-10.

SECONDARY OUTCOMES:
systemic analgesic administration times | 24 hour
  the first postoperative systemic analgesic administration time
frequency of systemic analgesic use | 24 hour
  the frequency of systemic analgesic use in the first 24 hours postoperatively
complications | 24 hour
  the complications related to the use of postoperative systemic analgesics and/or nerve block application

CONTACTS AND LOCATIONS:
Overall Officials: sebnem turk, Study Director — Sisli Hamidiye Etfal Training and Research Hospital
Locations (1):
- Sisli Hamidiye Etfal Training and Research Hospital, Şişli, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Samerchua A, Leurcharusmee P, Panichpichate K, Bunchungmongkol N, Wanvoharn M, Tepmalai K, Khorana J, Chantakhow S. A Prospective, randomized comparative study between ultrasound-guided posterior quadratus lumborum block and ultrasound-guided ilioinguinal/iliohypogastric nerve block for pediatric inguinal herniotomy. Paediatr Anaesth. 2020 Apr;30(4):498-505. doi: 10.1111/pan.13837. Epub 2020 Feb 21. PMID 32030845
- [Background] Priyadarshini K, Behera BK, Tripathy BB, Misra S. Ultrasound-guided transverse abdominis plane block, ilioinguinal/iliohypogastric nerve block, and quadratus lumborum block for elective open inguinal hernia repair in children: a randomized controlled trial. Reg Anesth Pain Med. 2022 Apr;47(4):217-221. doi: 10.1136/rapm-2021-103201. Epub 2022 Jan 17. PMID 35039439